CLINICAL TRIAL: NCT04502576
Title: Helmet Noninvasive Ventilation vs. High-flow Nasal Cannula in Moderate-to-severe Acute Hypoxemic Respiratory Failure: an Open Label, Pilot, Randomized Trial
Brief Title: Helmet Noninvasive Ventilation vs. High-flow Nasal Cannula in Moderate-to-severe Acute Hypoxemic Respiratory Failure
Acronym: HENIVOTpilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Università degli studi di Chieti (Unknown); Societa Italiana Anestesia Analgesia Rianimazione e Terapia Intensiva (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4443
Record Dates: First submitted 2020-08-03; First posted 2020-08-06 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2021-10

CONDITIONS: Respiratory Failure With Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-flow nasal cannula (Active Comparator): High-flow nasal cannula will be delivered with the Optiflow system. Initial set flow will be ≥ 50 /min and flows will be decreased in case of intolerance and/or according to patients' requirements: flows≥30 L/min will be mandatory in all enrolled patients. Humidification chamber (MR860, Fisher and Paykel healthcare, New Zealand) will be set at 37 °C or 34 °C according to patient's comfort. FiO2 will be titrated to obtain an SpO2≥92% and ≤98%.
  The treatment according to the assigned protocol will be continued until the patient requires endotracheal intubation or (in case of no intubation) up to ICU discharge. Weaning from high-flow will be considered as standardized criteria are met.
  Interventions: Device: Noninvasive respiratory support
- Helmet noninvasive ventilation (Experimental): Patients will receive continuous helmet pressure support ventilation for at least 16 hours/day the first 2 calendar days. Continuous noninvasive ventilation without interruptions will be strongly encouraged in the first 24 hours of treatment. The ventilator will be set in pressure support mode. Use of continuous positive airway pressure by flow generators and Venturi systems instead of pressure support ventilation will be allowed in case of shortage of ventilators. Maintenance of positive end-expiratory pressure ≥ 8-10 during the treatment is mandatory.
  After weaning and during any interruption from noninvasive ventilation, patients will undergo low-flow or high-flow oxygen, according to the decision of the attending physician.
  The treatment according to the assigned protocol will be continued until the patient requires endotracheal intubation or (in case of no intubation) up to ICU discharge.
  Interventions: Device: Noninvasive respiratory support

INTERVENTIONS:
Device: Noninvasive respiratory support — In both arms, the treatment according to the assigned protocol will be continued until the patient requires endotracheal intubation or (in case of no intubation) up to ICU discharge.
  Patients will have to undergo the allocated treatment within 1 hour from the moment of randomization and within 24 hours from admission in the intensive care unit

SUMMARY:
Helmet noninvasive ventilation and high-flow nasal cannula are novel tools for the first-line treatment of acute hypoxemic respiratory failure. Compared to face-mask noninvasive ventilation in randomized trials, both have improved clinical outcome of patients with moderate-to-severe hypoxemic respiratory failure.

As compared to high-flow nasal cannula, helmet noninvasive ventilation improves oxygenation, reduces inspiratory effort, respiratory rate and dyspnea. Whether these physiological benefits are translated into improved outcome remains to be established.

The investigators designed a randomized trial to establish whether first line treatment with Helmet noninvasive ventilation is capable of increasing the number of 28-day respiratory-support-free days, as compared to high-flow nasal cannula in patients with moderate-to-severe acute hypoxemic respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

Acute-onset respiratory distress or flue-related symptoms Moderate-to-severe hypoxemia (PaO2/FiO2<=200 mmHg) PaCO2<45 mmHg pH>7.30

Exclusion Criteria:

Need for urgent endo-tracheal intubation Exacerbation of asthma or chronic obstructive pulmonary disease Documented pneumothorax Clinical diagnosis of Cardiogenic pulmonary oedema Do-not-intubate order Altered neurological status that requires immediate intubation and/or making the patient uncooperative Thoracic or abdominal surgery in the previous 7 days Recent head surgery or anatomy that prevent the application of helmet or Optiflow to patient's face

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2021-01-10 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Respiratory-support free days within 28 days from randomization | 28 days
  The number of days in which patients did not receive any form of respiratory support (i.e. high-flow nasal cannula, noninvasive ventilation, invasive mechanical ventilation)

SECONDARY OUTCOMES:
Endotracheal intubation | 28 days
  The proportion of patients requiring endotracheal intubation in the two groups. The need for endotracheal intubation will be established with predefined criteria, which will be evaluated a posteriori by an independent adjudication committee
Invasive ventilation-free days within 28 days from randomization | 28 days
  The number of days in which patients did not receive invasive mechanical ventilation
Invasive ventilation-free days within 60 days from randomization | 60 days
  The number of days in which patients did not receive invasive mechanical ventilation
Oxygenation | 28 days
  The ratio of PaO2 to FiO2 will be measured 1, 6, 12, 24 hours after randomization and then once daily up to intensive care unit discharge
Carbon dioxide | 28 days
  PaCO2 will be measured 1, 6, 12, 24 hours after randomization and then once daily up to intensive care unit discharge
Dyspnea | 28 days
  Dyspnea will be evaluated through a visual analog scale (0-10, where 10 represents the most sever symptom) will be measured 1, 6, 12, 24 hours after randomization and then once daily up to intensive care unit discharge
Respiratory rate | 28 days
  Respiratory rate will be measured 1, 6, 12, 24 hours after randomization and then once daily up to intensive care unit discharge
In-intensive care unit mortality | 90 days
  Clinical outcome (dead/alive) at intensive care unit discharge
In-hospital mortality | 90 days
  Clinical outcome (dead/alive) at hospital discharge
90-day mortality | 90 days
  Clinical outcome (dead/alive) at 90 days after randomization
Quality of life after recovery | 1 year
  Quality of life in survivors, assessed by Short Form-36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Domenico Luca Grieco, MD, Principal Investigator — Fondazione Policlinico A. Gemelli IRCCS; Massimo Antonelli, MD, Study Director — Fondazione Policlinico A. Gemelli IRCCS
Locations (5):
- Italy (5):
  - Policlinico di Sant'Orsola, Alma Mater Studiorum-Università di Bologna, Bologna
  - SS. Annunziata Hospital, Gabriele d'Annunzio University of Chieti-Pescara, Chieti
  - Azienda Ospedaliera-Universitaria Arcispedale Sant'Anna, University of Ferrara, Ferrara
  - Infermi Hospital, Rimini
  - Fondazione Policlinico Universitaro A. Gemelli IRCCS, Rome

IPD SHARING:
Plan to Share IPD: Undecided
Data will be made available upon a reasonable request

REFERENCES:
- [Derived] Michi T, Mattana C, Menga LS, Bocci MG, Cesarano M, Rosa T, Gualano MR, Montomoli J, Spadaro S, Tosato M, Rota E, Landi F, Cutuli SL, Tanzarella ES, Pintaudi G, Piervincenzi E, Bello G, Tonetti T, Rucci P, De Pascale G, Maggiore SM, Grieco DL, Conti G, Antonelli M; Gemelli COVID-ICU study group. Long-term outcome of COVID-19 patients treated with helmet noninvasive ventilation vs. high-flow nasal oxygen: a randomized trial. J Intensive Care. 2023 May 19;11(1):21. doi: 10.1186/s40560-023-00669-0. PMID 37208787
- [Derived] Grieco DL, Menga LS, Cesarano M, Rosa T, Spadaro S, Bitondo MM, Montomoli J, Falo G, Tonetti T, Cutuli SL, Pintaudi G, Tanzarella ES, Piervincenzi E, Bongiovanni F, Dell'Anna AM, Delle Cese L, Berardi C, Carelli S, Bocci MG, Montini L, Bello G, Natalini D, De Pascale G, Velardo M, Volta CA, Ranieri VM, Conti G, Maggiore SM, Antonelli M; COVID-ICU Gemelli Study Group. Effect of Helmet Noninvasive Ventilation vs High-Flow Nasal Oxygen on Days Free of Respiratory Support in Patients With COVID-19 and Moderate to Severe Hypoxemic Respiratory Failure: The HENIVOT Randomized Clinical Trial. JAMA. 2021 May 4;325(17):1731-1743. doi: 10.1001/jama.2021.4682. PMID 33764378